CLINICAL TRIAL: NCT00491348
Title: Effects of Duloxetine on Pathological Worry in Patients With Generalized Anxiety Disorder: A fMRI Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of MRI mode
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Mei-Chih Tseng/Attending psychiatrist, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 950508
Record Dates: First submitted 2007-06-23; First posted 2007-06-26 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Worry; Anxiety
Keywords: Generalized anxiety disorder; fMRI; Worry
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: duloxetine hydrochloride — duloxetine 30 mg QD, may titrate to 30 mg BID, and maintain the dosage for 6 weeks
  Other Names: Cymbalta

SUMMARY:
(1) to compare the differences of neural activation of pathological worry between pre-treatment GAD patients and normal subjects; (2) to measure the differences of brain activation on worry in GAD patients before and after duloxetine treatment

DETAILED DESCRIPTION:
The study will recruit 20 GAD patients and 20 healthy controls. Both patients and controls receive a medical and psychiatric screening procedure at visit 1 and are asked to complete three self-rating questionnaires and one health questionnaire at visit 1. All qualified participants will receive functional magnetic resonance imaging (fMRI) at baseline.

The patients will begin treatment with duloxetine 30 mg/day at visit 2 and will be titrated to 60 mg/day at visit 3 (2 week since drug dispensed). The dosage will be maintained on 60 mg/day for 6 more weeks. During the period, the patients will receive periodic evaluations at visit 2 (0 week drug dispensed), 3 (2 week since drug dispensed), 4 (4 weeks since drug dispensed), and 5 (8 weeks since drug dispensed). The patients will receive fMRI examination at baseline and at the end of the 8-week treatment.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria of generalized anxiety disorders with moderate degree
* Participants above 18 years old

Exclusion Criteria:

* Major depression
* Panic disorder
* Obsessive-compulsive disorder
* Post-traumatic disorder
* Eating disorders
* Psychotic disorders; and
* Alcohol or other substance use disorders
* Neurological disease
* Cardio-vascular disease
* Respiratory disease
* Head trauma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
difference of brain activation on worry | two months

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Chih Tseng, MD, Study Director — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan